CLINICAL TRIAL: NCT03279016
Title: Diagnosis of Temporomandibular Joint Arthritic Disease Using Arthroscopic Guided Synovial Biopsies
Brief Title: Arthroscopic Guided Synovial Biopsies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Adel EISSA, doctor, Cairo University
Other Study IDs: CEBD-CU-2017-08-28
Record Dates: First submitted 2017-08-31; First posted 2017-09-12 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Temporomandibular Arthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To detect accuracy of serology in diagnosis of temporomandibular joint arthritis.

DETAILED DESCRIPTION:
According to a search of previously published studies on accuracy of serology no sensitivity or specificity data was found regarding accurate detection of arthritis through serology, hence the aim of this study is to detect accuracy of serology in diagnosis of temporomandibular joint arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from TEMPOROMANDIBULAR JOINT ARTHRITIS.
* Patients should be free from any systemic disease that may affect normal healing and predictable outcome.
* Patients who will agree to the consent

Exclusion Criteria:

* Patients with any systemic disease that may affect normal healing.
* Pregnant females.
* Patients with acute infection.
* Patients with bony ankyloses.
* Patients with risk of tumor dissemination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient complaing from arthritis symptoms,an diagnosed as arthritic patient with MRI
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
accuracy of serology | 2 years
  To determine the sensitivity or specificity of serology in diagnosis of temporomandibular joint arthritis

SECONDARY OUTCOMES:
Rheumatoid factor | 2 years
  To be measured in a blood sample with (IU/mL) unit as The normal reference range for RF is less than 15 IU/mL
C-reactive protein | 2 years
  To be measured in a blood sample with (mg/dL) unit where Normal CRP levels are below 3.0 mg/dL.
Anti-Cyclic Citrullinated Peptide | 2 years
  To be measured in a blood sample with (titre-AU)
ANA | 2 years
  To be measured in a blood sample with binary outcome (positive or negative)
HLA-B27 | 2 years
  To be measured in a blood sample with binary outcome (positive or negative)
Cellular population- type | 2 years
  Presence of inflammatory cells infiltrate at the synovial membrane biopsy :
  - type of cells
Cellular population- number of cells | 2 years
  Presence of inflammatory cells infiltrate at the synovial membrane biopsy:
  - mean number of cells

CONTACTS AND LOCATIONS:
Overall Officials: sameh mekhaimer, professor, Study Director — professor of oral and maxillofacial surgery,faculty of oral and dental medicine,Cairo university
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided